CLINICAL TRIAL: NCT02823223
Title: A Multi-center, Prospective, Randomized, Controlled Trial of Endobronchial Valve Therapy vs. Standard of Care in Heterogeneous Emphysema
Brief Title: Endobronchial Valve in Patients With Heterogeneous Emphysema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Liang_An, MD,PHD, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2016-026-01
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
Keywords: Endobronchial Valve
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELVR with Endobronchial Valves (Experimental): Patients will have ELVR (Endoscopic Lung Volume Reduction) with Endobronchial Valves (Zephyr valve) inserted into the target lobe of the lung with the aim of complete lobar exclusion.
  Interventions: Device: Zephyr endobronchial valve placement
- Standard of Care (No Intervention): Patients will receive optimal drug therapy and medical management according to clinical practice

INTERVENTIONS:
Device: Zephyr endobronchial valve placement — Patients will have ELVR (Endoscopic Lung Volume Reduction) with Zephyr valve inserted into the target lobe of the lung with the aim of complete lobar exclusion.
  Arms: ELVR with Endobronchial Valves

SUMMARY:
To compare the clinical outcomes of Endoscopic Lung Volume Reduction using Pulmonx Zephyr Endobronchial Valve (EBV) vs. Standard of Care (SoC) in the treatment of heterogeneous emphysema patients in a controlled trial design setting.

DETAILED DESCRIPTION:
The aim of this prospective, randomized, controlled, one-way crossover study is to assess and compare the efficacy of the Zephyr endobronchial valves vs. Standard of Care (SoC) in patients suffering from COPD with Heterogeneous Emphysema. Patients will be followed up for 6 months after randomization. Patients in the SoC arm will crossover to the EBV treatment arm after the 6-month visit and will be followed up for 6 additional months.The primary objective is the variation of FEV1 between baseline and 3-month follow-up visit. The secondary objectives will evaluate quality of life, exercise capacity, dyspnea (including BODE index) changes, target lobe volume reduction, as well as safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Consent form signed
* Heterogeneous emphysema on Chest CT Scanner
* Intact interlobar fissures adjacent to the target lobe on Chest CT or collateral ventilation negative in the target lobe by Chartis assessment
* Post bronchodilator Forced expiratory volume in 1 second (FEV1) < 50% predicted
* Total Lung Capacity > 100% predicted
* Residual Volume > 150% predicted
* PaO2 > 45mmHg
* Post rehabilitation 6 minute walk test > 140m
* No COPD exacerbation for at least 6 weeks
* Stopped cigarette smoking for more than 3 months

Exclusion Criteria:

* Contraindication to bronchoscopy
* Tuberculosis, pleural effusion, or clinically significant bronchiectasis
* Lung carcinoma or pulmonary nodule on CT scan requiring Chest CT scan follow-up
* Active pulmonary infection
* Prior lung transplant, LVRS, median sternotomy, bullectomy or lobectomy
* Any extrapulmonary diseases compromising survival or evaluation within the protocol (severe cardiac disease, severe renal insufficiency, cancer…)
* Inclusion in an other study assessing respiratory treatments
* Pregnant or lactating woman

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change in Forced Expiratory Volume in 1 s (FEV1) | At baseline and after 3 months

SECONDARY OUTCOMES:
Percentage change in Forced Expiratory Volume in 1 s (FEV1) | At baseline and after 6 months
Comparison of the FEV1 using 15% Percentage change as cut-off for clinically significant change | At baseline and after 3, 6 months
Change in Residual Volume (RV) | At baseline and after 3, 6 months
Change in Total Lung Capacity (TLC) | At baseline and after 3, 6 months
Change in FEV1/FVC ratio | At baseline and after 3, 6 months
Change in St George's Respiratory Questionnaire | At baseline and after 3, 6 months
Change in 6-Min Walk Test | At baseline and after 3, 6 months
Change in BODE index | At baseline and after 3, 6 months
Change in mMRC score | At baseline and after 3, 6 months
Adverse Events and Serious Adverse Events | At each visits
  AEs: Type, incidence, severity, seriousness and relationship to study medications of adverse events (AE) (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE 4.0]

CONTACTS AND LOCATIONS:
Overall Officials: Liang_an Chen, MD, phD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Because of personal privacy, the research-related individual participant data do not intend for public sharing.